CLINICAL TRIAL: NCT01451593
Title: A Phase II Double Blind, Randomized, Placebo Controlled Trial of Neuroprotection With Phenytoin in Acute Optic Neuritis
Brief Title: Neuroprotection With Phenytoin in Optic Neuritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Multiple Sclerosis Society (Other); Multiple Sclerosis Society of Great Britain and Northern Ireland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCL/11/0083
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Optic Neuritis; Multiple Sclerosis
Keywords: Optic neuritis; Multiple sclerosis; Retinal nerve fibre layer; Axonal loss; Neuroprotection; Phenytoin; MRI; Optical coherence tomography; Sodium Channel Blockers
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis | interventions — Phenytoin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- phenytoin (Experimental): active arm of trial 1:1 allocation active versus placebo
  Interventions: Drug: Phenytoin
- placebo (Placebo Comparator): 1:1 allocation active versus placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Phenytoin — Phenytoin will be loaded using at total dose of 15mg/kg (rounded to the nearest 100mg) divided into three equal doses given once daily for 3 days.This will be followed by a daily maintenance dose of 4mg/kg once a day (rounded up to the nearest 50mg, with a maximum dose of 300mg)for 13 weeks.Phenytoin levels will be taken at 1 and 3 months.
  Other Names: Phenytoin sodium; Epanutin (Flynn Pharma)
  Arms: phenytoin
Drug: Placebo — placebo identical in appearance to active IMP (phenytoin)
  Arms: placebo

SUMMARY:
Optic neuritis is caused by inflammation of the optic nerve and causes loss of vision in the affected eye. It is often associated with multiple sclerosis. Loss of vision after an attack of optic neuritis is caused by damage to the nerve fibres in the optic nerve. There are a number of factors that contribute to nerve fibre damage including increased levels of sodium within them, so blocking sodium entry could help to protect them against damage.

The purpose of this study is determine whether phenytoin (which blocks sodium entry into cells) can protect against loss of nerve fibres and prevent loss of vision after optic neuritis.

DETAILED DESCRIPTION:
Demyelinating optic neuritis is the most common cause of acute reversible visual loss in young adults of Northern European Origin. There is a strong association with multiple sclerosis and up to 75% of British adults with acute clinically isolated optic neuritis go on to develop MS during long term follow up. Equally, 70% of MS patients have clinical evidence if optic nerve involvement during the course of their illness.

The pathology of the acute inflammatory lesion is comparable to the plaques found elsewhere in the CNS in MS. The retina and optic nerve therefore represent a discrete compartment of the CNS affected by the disease process that can be easily studied using a combination of clinical, electrophysiological and imaging techniques.

There is good evidence that axonal and neuronal degeneration are the primary pathological processes leading to irreversible disability in MS. Experimental models have demonstrated numerous mechanisms of axonal loss including adaptive changes in the demyelinated axonal membrane, in particular increased density of sodium channels leading to increased concentrations of intraaxonal sodium ions. Partial blockade of voltage gated sodium channels with drugs such as phenytoin has been shown to be neuroprotective in several experimental models of inflammatory axonal injury.

The retinal nerve fibre layer is unique in the CNS in that it is not myelinated and therefore is an ideal biomarker for the processes of neurodegeneration and neuroprotection.

Imaging of the retinal nerve fibre layer using optical coherence tomography and of the optic nerve using MRI both demonstrate that acute optic neuritis is associated with significant volume loss, and this correlates well with impaired visual function.

The primary aim of this trial is to assess whether sodium channel blockade with phenytoin has a neuroprotective effect on axonal loss after an attack of acute demyelinating optic neuritis. Secondary aims are to assess whether phenytoin improves visual outcome and remyelination and to assess the safety of the treatment.

90 patients with acute optic neuritis will be recruited into a double blind placebo controlled trial in which patients will be randomly allocated to receive either phenytoin or placebo for 3 months. Recruitment will take place at two trial sites in Sheffield and London. The trial is powered to detect a 50% beneficial effect on the primary outcome measure. Outcome will be measured at entry and after 6 months.Bias will be minimized by blinding assessing physicians and patients using active and placebo treatment of identical appearance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute optic neuritis
* Visual acuity in affected eye ≤ 6/12
* Corrected vision in normal eye ≥ 6/6
* No history of optic neuritis or other ocular disease in either eye
* ≤ 14 days since onset of visual loss

Exclusion Criteria:

* Contraindication or known allergy to Phenytoin
* Contraindication to MRI
* Use of a calcium channel or sodium channel blocker in the past 2 months
* Corticosteroid use in the past 2 months
* Tysabri infusion in the past 3 months
* MS with major temperature dependent disability
* Relapsing remitting MS of greater than 10 yrs duration or EDSS>3
* Pregnancy
* Breast Feeding
* Significant cardiac, renal or liver abnormalities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean Retinal nerve fibre layer thickness | Measured at entry and after 6 months
  The primary comparison will estimate active versus placebo mean retinal nerve fibre layer thickness of the retinal nerve fibre layer after 6 months, adjusted for the corresponding baseline measurement in the unaffected eye.

SECONDARY OUTCOMES:
Visual function | Measured at entry and 6 months
  logMAR visual acuity, low contrast sensitvity using 1.25% and 2.5% sloan charts and colour vision using Farnsworth-Munsell 100 Hue test.
Visual evoked potentials | Measured at entry (or within 4 weeks) and after 6 months
  Measurement of latency and amplitude will be performed. Axonal protection with phenytoin may enable axons to survive long enough to undergo remyelination. VEPS will give independent estimates of remyelination in the optic nerve.
Optic nerve and brain MRI | Brain MRI will be performed at entry(or within 4 weeks) Optic nerve MRI will be performed at entry (or within 4 weeks) and after 6 months
  Brain MRI to detect demyelinating lesions that can be used in considering the prognosis for or diagnosis of multiple sclerosis using McDonald criteria.
  Optic nerve MRI - The following sequences will be performed:
  1. Fat sat T2 coronal-oblique to visualize the symptomatic lesion and obtain optic nerve area measurements.
  2. 3D gradient echo magnetization transfer sequence MTR to obtain measures of optic nerve myelination.
  3. Diffusion tensor imaging to obtain axial and radial diffusivity metrics of the optic nerve to determine axonal integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Raju Kapoor, DM FRCP, Principal Investigator — Institute of Neurology, University College London
Locations (2):
- United Kingdom (2):
  - National Hospital for Neurology and Neurosurgery, London
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Kodali S, Bianchi A, Raftopoulos R, Moccia M, Malladi AP, Yiannakas MC, Fugger M, Samson RS, Wheeler-Kingshott CAM, Koltzenburg M, Prados F, Hickman S, Kapoor R, Toosy AT. Effects of Phenytoin on the Retinal Ganglion Cell-Inner Plexiform Layer in Acute Optic Neuritis: Analysis of a Phase II Randomized Trial. Neurology. 2025 Oct 21;105(8):e213951. doi: 10.1212/WNL.0000000000213951. Epub 2025 Sep 25. PMID 40997284
- [Derived] Raftopoulos R, Hickman SJ, Toosy A, Sharrack B, Mallik S, Paling D, Altmann DR, Yiannakas MC, Malladi P, Sheridan R, Sarrigiannis PG, Hoggard N, Koltzenburg M, Gandini Wheeler-Kingshott CA, Schmierer K, Giovannoni G, Miller DH, Kapoor R. Phenytoin for neuroprotection in patients with acute optic neuritis: a randomised, placebo-controlled, phase 2 trial. Lancet Neurol. 2016 Mar;15(3):259-69. doi: 10.1016/S1474-4422(16)00004-1. Epub 2016 Jan 26. PMID 26822749
- [Derived] Counihan TJ, Duignan JA, Gormley G, Saidha S, Dooley C, Newell J. Does long-term partial sodium channel blockade alter disease progression in MS? Evidence from a retrospective study. Ir J Med Sci. 2014 Mar;183(1):117-21. doi: 10.1007/s11845-013-1042-7. Epub 2013 Nov 28. PMID 24287594